CLINICAL TRIAL: NCT03669224
Title: Marginal Integrity of Resin Composite Restoration With & Without Surface Pretreatment by Gold & Silver Nanoparticles Versus Chlorhexidine in Class II Cavities Randomized Controlled Trial
Brief Title: Effect of Nano Care Gold on Marginal Integrity of Resin Composite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Abd El-Fattah Mohammed, Assistant Lecturer of Conservative Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-04
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Caries Class Ii
Keywords: marginal adptation; marginal staining; post operative sensitivity; recurrent caries
MeSH Terms: interventions — Silver; Chlorhexidine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nano Care Gold (Experimental): Silver and Gold nano particles suspended in 70 % isopropyl alcohol. It will be used for cavity pre-treatment. This arm will be compared with no intervention (negative control).
  Interventions: Other: Nano Care Gold; Other: No intervention
- Chlorhexidine (Active Comparator): 2% chlorhexidine gluconate solution will be applied to prepared cavity followed by adhesive system then resin composite. This arm will be compared with no intervention (negative control).
  Interventions: Other: No intervention; Other: Chlorhexidine

INTERVENTIONS:
Other: Nano Care Gold — Mixture of Gold and Silver nano particles suspended in 70 % Isopropyl alcohol. This group will be compared with no intervention group.
  Other Names: Silver and Gold nano particles
  Arms: Nano Care Gold
Other: No intervention — No intervention will be applied in this group. It will be the negative comparator. In this group only the standard of care will be applied, which means the steps will be cavity preparation followed by adhesive system then resin composite without any surface pre-treatment
  Other Names: Negative control
Other: Chlorhexidine — 2 % chlorhexidine gluconate. This group will be compared with no intervention group.
  Other Names: chlorhexidine gluconate
  Arms: Chlorhexidine

SUMMARY:
The aim of this study to detect the effect of Nano Care Gold on marginal integrity of resin composite restoration

DETAILED DESCRIPTION:
This study will be divided into 3 groups (control, Nano Care Gold, Chlorhexidine). Both materials will be used as a surface pre-treatment. Their effect on marginal integrity will be evaluated through evaluation of marginal adaptation, marginal staining, post-operative sensitivity. The follow up period is one year

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with at least two class II cavities (2) 17-50 years old (3) Males or females (4) Good or hygiene (5) Good general health (6) Cooperative patients (7) Subjects who signed the informed consent

Exclusion Criteria:

1. Patients younger than 17 years or older than 50 years old
2. Pregnant females
3. Disabilities
4. Systemic disease or severe medical complications
5. Heavy smoking
6. Lack of compliance

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | 1 year
  It will be measured by FDI probe and Digora x-ray machine. FDI Scoring system (categorical) 5 steps(3 accepted, 2 unaccepted) will be used to evaluate the outcome of measuring device

SECONDARY OUTCOMES:
Marginal staining | 1 year
  Visual inspection and Photographs will be used to measure the outcome. FDI Scoring system(categorical) 5 steps(3 accepted, 2 unaccepted) will be used to evaluate the outcome
Post operative sensitivity | 1 year
  A blast of cold air will be used to evaluate the restoration. FDI Scoring system(categorical) 5 steps(3 accepted, 2 unaccepted) will be used to determine the restoration fit in which category.

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Abd El-Fattah Mohammed Nemtallah, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Effect of Gold and Silver nano particles on marginal adaptation of resin composite